CLINICAL TRIAL: NCT04411823
Title: Prediction of Post-laparoscopic Sleeve Gastrectomy Gastroesophageal Reflux Disease With an Endolumenal Functional Lumen Imaging Probe (EndoFLIP)
Brief Title: Post-sleeve Gastrectomy Gastroesophageal Reflux Disease Prediction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Omar Ghanem, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-000348
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Gastroesophageal Reflux; Sleeve Gastrectomy; Bariatric Surgery Complication
Keywords: Gastroesophageal Reflux; Sleeve gastrectomy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention arm (Experimental): Undergo an upper endoscopy with EndoFLIP at baseline before sleeve gastrectomy
  Interventions: Device: EndoFLIP measurement

INTERVENTIONS:
Device: EndoFLIP measurement — EndoFLIP device can measure gastroesophageal junction distensibility index and esophageal contractile pattern under FDA cleared indication. It is performed during endoscopy.

SUMMARY:
Researchers are trying to identify predictors for gastroesophageal reflux disease after sleeve gastrectomy.

DETAILED DESCRIPTION:
Subjects will undergo an upper endoscopy with EndoFLIP before sleeve gastrectomy to measure parameters from endoscopy and EndoFLIP device to develop a prediction model for post-operative gastroesophageal reflux disease. Subjects will undergo a repeat upper endoscopy with EndoFLIP at 6 months if an upper endoscopy is clinically indicated after surgery and complete questionnaires during follow-ups up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years
* BMI 30 or greater kg/m2
* Participants can give a consent to the procedure
* Participants have no contraindications to LSG (gastric ulceration)

Exclusion Criteria:

* Participants who have LA grade C or D esophagitis, Barrett mucosa or peptic stricture.
* Patients who have evidence of a major motility abnormality defined by the Chicago classification version 3.0 (achalasia, absent contractility, esophagogastric junction outflow obstruction, distal esophageal spasm, or hypertensive peristalsis)
* Patients with hiatal hernia > 3 cm
* Patients with previous esophageal or stomach surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Worsening or new-onset gastroesophageal reflux disease | Baseline, 6 months, and 5 years
  Determined by the change in the GERD-Health Related Quality of Life questionnaire score with questions individually scored on a scale of 0-5, combined to determine a total score range of 0-75 where a higher score indicates worse quality of life and increased score would indicate new or worsening GERD.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ghanem, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Orlando Health, Orlando, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials